CLINICAL TRIAL: NCT01390844
Title: Safety and Efficacy of Boceprevir in Combination With Peginterferon Plus Ribavirin for Treatment of Asia Pacific Subjects With Chronic Hepatitis C Genotype 1 Who Failed Prior Treatment With Pegylated Interferon Plus Ribavirin
Brief Title: Safety and Efficacy of Boceprevir in Asia Pacific Participants With Chronic Hepatitis C Genotype 1 (P07063)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P07063; 2007-005151-42 (EudraCT Number); 3034-033 (Other: Merck study number); CTRI/2012/04/002540 (Registry Identifier: CTRI)
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Results first posted 2016-06-28 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Boceprevir (Experimental): PEG + RBV for 4 weeks followed by BOC + PEG + RBV for 32 weeks. At the Treatment Week 36 visit, participants with undetectable HCV-RNA at Treatment Weeks 8 and 12 will proceed to 36 weeks of post-treatment follow-up. Participants with detectable HCV-RNA at Treatment Week 8 and undetectable HCV-RNA at Treatment Week 12 will continue on BOC + PEG + RBV until Treatment Week 36, receive placebo + PEG + RBV until Treatment Week 48, and then proceed to 24 weeks of post-treatment follow-up. Participants with any HCV-RNA result at Treatment Week 8 and detectable HCV-RNA at Treatment Week 12 will discontinue treatment and proceed to 24 weeks of post-treatment follow-up.
  Interventions: Drug: Boceprevir (BOC); Drug: Placebo to boceprevir; Drug: Peginterferon alfa-2b (PEG); Drug: Ribavirin (RBV)
- Control (Active Comparator): PEG + RBV for 4 weeks followed by BOC placebo + PEG + RBV for 44 weeks. Participants with undetectable HCV-RNA at Treatment Week 12 and at subsequent assays will continue on placebo + PEG + RBV through Treatment Week 48 and proceed to 24 weeks of post-treatment follow-up. Participants with detectable HCV-RNA at Treatment Week 12 may roll over to Cross-Over BOC treatment beginning with Treatment Week 14.
  Interventions: Drug: Placebo to boceprevir; Drug: Peginterferon alfa-2b (PEG); Drug: Ribavirin (RBV); Drug: Cross-Over Boceprevir Treatment

INTERVENTIONS:
Drug: Boceprevir (BOC) — 200 mg capsules, 800 mg three times daily by mouth
  Other Names: SCH 503034; Victrelis
  Arms: Boceprevir
Drug: Placebo to boceprevir — 200 mg placebo capsules, 800 mg three times daily by mouth
Drug: Peginterferon alfa-2b (PEG) — 1.5 mcg/kg/week subcutaneously
  Other Names: PegIntron; SCH 054031; Redipen
Drug: Ribavirin (RBV) — 200 mg capsules, weight-based dosing 800 to 1400 mg/day by mouth divided twice daily
  Other Names: Rebetol; SCH 018908
Drug: Cross-Over Boceprevir Treatment — At Treatment Week 14, participants in the Placebo group with detectable HCV-RNA at Treatment Week 12 have the option to add boceprevir 800 mg three times daily to the PEG + RBV regimen for up to 32 weeks.
  Other Names: SCH 503034; Victrelis
  Arms: Control

SUMMARY:
This study will assess the efficacy of boceprevir (BOC) in combination with PegIntron (pegylated interferon alfa-2b) (PEG) and ribavirin (RBV) in response guided therapy compared to the efficacy of standard-of-care therapy alone in adult subjects with chronic hepatitis C (CHC) genotype 1 who failed prior treatment with pegylated interferon and RBV in the Asia Pacific population. The primary hypothesis is that the proportion of participants achieving sustained virologic response in the experimental therapy regimen (BOC/PEG+RBV) is superior to that in the control arm (Placebo/PEG+RBV), in the Full Analysis Set (FAS) population.

ELIGIBILITY:
Inclusion Criteria:

* Previously documented CHC genotype 1 infection. Other or mixed genotypes are not eligible.
* Liver biopsy with histology consistent with CHC and no other etiology.
* Participants with cirrhosis must have an ultrasound/imaging study within 6 months of screening (or between screening and Day 1) with no findings suspicious for hepatocellular carcinoma
* Failed previous treatment (of at least 12 weeks) with pegylated interferon (alfa-2a or alfa-2b) plus RBV
* Weight between 40 kg and 125 kg, inclusive
* Of 'local' ancestral descent
* Sexually active males and females of child-bearing potential must agree to use a medically accepted method of contraception

Exclusion Criteria:

* Co-infected with the human immunodeficiency virus (HIV) or hepatitis B virus.
* Required discontinuation of previous interferon or RBV regimen for an adverse event considered to be possibly or probably related to RBV and/or interferon.
* Treatment with RBV within 90 days and any interferon-alpha within 1 month prior to screening.
* Treatment for hepatitis C with any investigational medication or prior treatment with herbal remedies with known hepatotoxicity.
* Treatment with any investigational drug or participation in any interventional clinical trial within 30 days of the screening visit.
* Evidence of decompensated liver disease including, but not limited to, a history or presence of clinical ascites, bleeding varices, or hepatic encephalopathy.
* Diabetes and/or hypertension with clinically significant ocular examination findings.
* Any condition the could interfere with participation in and completion of the trial.
* Evidence of active or suspected malignancy, or history of malignancy within the last 5 years (except adequately treatment carcinoma in situ and basal cell carcinoma of the skin).
* Pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2011-10-21 (Actual); Primary Completion 2015-06-19 (Actual); Study Completion 2015-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants in an Asia Pacific population with chronic Hepatitis C (CHC) genotype 1 who have failed prior treatment with pegylated interferon and ribavirin (PR) were selected to participate in this study.
Pre-assignment Details: Of 282 participants randomized and treated, 269 participants followed Good Clinical Practice (GCP); 13 participants did not follow GCP.
Groups:
- Boceprevir - Korea+Taiwan: PegIntron (pegylated interferon alfa-2b) (PEG) + ribavirin (RBV) for 4 weeks followed by boceprevir (BOC) + PEG + RBV for 32 weeks. At the Treatment Week 36 visit, participants with undetectable hepatitis C virus ribonucleic acid (HCV-RNA) at Treatment Weeks 8 and 12 will proceed to 36 weeks of post-treatment follow-up. Participants with detectable HCV-RNA at Treatment Week 8 and undetectable HCV-RNA at Treatment Week 12 will continue on BOC + PEG + RBV until Treatment Week 36, receive placebo + PEG + RBV until Treatment Week 48, and then proceed to 24 weeks of post-treatment follow-up. Participants with any HCV-RNA result at Treatment Week 8 and detectable HCV-RNA at Treatment Week 12 will discontinue treatment and proceed to 24 weeks of post-treatment follow-up.
- Control - Korea+Taiwan; Control - India: PEG + RBV for 4 weeks followed by BOC placebo + PEG + RBV for 44 weeks. Participants with undetectable HCV-RNA at Treatment Week 12 and at all subsequent assays will continue on placebo + PEG + RBV through Treatment Week 48 and proceed to 24 weeks of post-treatment follow-up. Participants with detectable HCV-RNA at Treatment Week 12 may roll over to Cross-Over BOC treatment beginning with Treatment Week 14.
- Boceprevir - India: PEG + RBV for 4 weeks followed by BOC + PEG + RBV for 32 weeks. At the Treatment Week 36 visit, participants with undetectable HCV-RNA at Treatment Weeks 8 and 12 will proceed to 36 weeks of post-treatment follow-up. Participants with detectable HCV-RNA at Treatment Week 8 and undetectable HCV-RNA at Treatment Week 12 will continue on BOC + PEG + RBV until Treatment Week 36, receive placebo + PEG + RBV until Treatment Week 48, and then proceed to 24 weeks of post-treatment follow-up. Participants with any HCV-RNA result at Treatment Week 8 and detectable HCV-RNA at Treatment Week 12 will discontinue treatment and proceed to 24 weeks of post-treatment follow-up.
Period: Treatment Phase
Arm/Group | Boceprevir - Korea+Taiwan | Control - Korea+Taiwan | Boceprevir - India | Control - India
Started | 133 | 65 | 57 | 27
Followed Good Clinical Practice (GCP) | 133 | 65 | 47 | 24
Completed | 93 | 37 | 26 | 8
Not Completed | 40 | 28 | 31 | 19
Not completed — Adverse Event | 12 | 2 | 3 | 2
Not completed — Treatment Failure | 23 | 25 | 10 | 13
Not completed — Non-Medical Reasons | 5 | 1 | 8 | 1
Not completed — Non-GCP Compliant | 0 | 0 | 10 | 3
Period: Follow-Up Phase
Arm/Group | Boceprevir - Korea+Taiwan | Control - Korea+Taiwan | Boceprevir - India | Control - India
Started | 93 | 37 | 26 | 8
Completed | 92 | 36 | 25 | 8
Not Completed | 1 | 1 | 1 | 0
Not completed — Non-Medical Reasons | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All Participants Randomized
Groups:
- Boceprevir - Korea+Taiwan; Boceprevir - India: PEG + RBV for 4 weeks followed by BOC + PEG + RBV for 32 weeks. At the Treatment Week 36 visit, participants with undetectable HCV-RNA at Treatment Weeks 8 and 12 will proceed to 36 weeks of post-treatment follow-up. Participants with detectable HCV-RNA at Treatment Week 8 and undetectable HCV-RNA at Treatment Week 12 will continue on BOC + PEG + RBV until Treatment Week 36, receive placebo + PEG + RBV until Treatment Week 48, and then proceed to 24 weeks of post-treatment follow-up. Participants with any HCV-RNA result at Treatment Week 8 and detectable HCV-RNA at Treatment Week 12 will discontinue treatment and proceed to 24 weeks of post-treatment follow-up.
- Total: Total of all reporting groups
Arm/Group | Boceprevir - Korea+Taiwan | Control - Korea+Taiwan | Boceprevir - India | Control - India | Total
Number analyzed (Participants) | 133 | 65 | 57 | 27 | 282
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.0 (10.15) | 52.4 (9.80) | 47.9 (9.83) | 45.2 (12.27) | 51.6 (10.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 28 | 18 | 5 | 99
  Male | 85 | 37 | 39 | 22 | 183

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Korea and Taiwan With Sustained Virologic Response (SVR) at Follow-Up Week 24 - Full Analysis Set (FAS) Population
Description: SVR is defined as undetectable plasma HCV-RNA at Follow-up Week (FW) 24. If FW24 is missing and other HCV-RNA values after FW24 are available, the last available value would be used for FW24. The last observation carried forward (LOCF) method was used to impute missing values; if a participant is missing at and after FW24 and has FW12 data, then FW12 data will be carried forward to FW24. Cross-over participants are considered as non-responders in SVR.
Time Frame: Follow-up Week 24
Population: FAS - population includes all randomized participants who received at least one (1) dose of any study medication (i.e., PEG, RBV, or BOC).
Measure: Number; unit: Percentage of Participants
Arm/Group | Boceprevir - Korea+Taiwan | Control - Korea+Taiwan
Number analyzed (Participants) | 133 | 65
Percentage of Participants | 60.90 | 26.15
Statistical Analysis 1: Comparison: Boceprevir - Korea+Taiwan vs Control - Korea+Taiwan; Between-Group Comparison; Test type: Superiority or Other; p < 0.0001, Miettinen and Numinen; Difference in Percentage = 34.63, 95% CI 2-sided [20.24 to 47.18]

2. Primary Outcome: Percentage of Participants in India With SVR at Follow-Up Week 24 - FAS Population
Description: SVR is defined as undetectable plasma HCV-RNA at FW24. If FW24 is missing and other HCV-RNA values after FW24 are available, the last available value would be used for FW24. The LOCF method was used to impute missing values; if a participant is missing at and after FW24 and has FW12 data, then FW12 data will be carried forward to FW24. Cross-over participants are considered as non-responders in SVR.
Time Frame: Follow-up Week 24
Population: FAS - population includes all randomized participants who received at least one (1) dose of any study medication (i.e., PEG, RBV, or BOC); participants who did not demonstrate GCP compliance were excluded from analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Boceprevir - India | Control - India
Number analyzed (Participants) | 47 | 24
Percentage of Participants | 53.19 | 20.83
Statistical Analysis 1: Comparison: Boceprevir - India vs Control - India; Between-Group Comparison; Test type: Superiority or Other; p = 0.0063, Miettinen and Numinen; Difference in Percentage = 33.83, 95% CI 2-sided [10.15 to 52.18]

3. Secondary Outcome: Percentage of Participants in Korea and Taiwan With SVR at Follow-Up Week 24 - Modified Intent-to-Treat (mITT) Population
Description: as for outcome 2
Time Frame: Follow-up Week 24
Population: mITT - population includes all randomized participants who received at least one (1) dose of experimental study drug (i.e., BOC for the Experimental Arm or placebo for the Control Arm).
Measure: Number; unit: Percentage of Participants
Arm/Group | Boceprevir - Korea+Taiwan | Control - Korea+Taiwan
Number analyzed (Participants) | 131 | 64
Percentage of Participants | 61.83 | 26.56
Statistical Analysis 1: Comparison: Boceprevir - Korea+Taiwan vs Control - Korea+Taiwan; Between-Group Comparison; Test type: Superiority or Other; p < 0.0001, Miettinen and Numinen; Difference in Percentage = 35.05, 95% CI 2-sided [20.51 to 47.72]

4. Secondary Outcome: Percentage of Participants in India With SVR at Follow-Up Week 24 - mITT Population
Description: as for outcome 2
Time Frame: Follow-up Week 24
Population: mITT - population includes all randomized participants who received at least one (1) dose of experimental study drug (i.e., BOC for the Experimental Arm or placebo for the Control Arm); participants who did not demonstrate GCP compliance were excluded from analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Boceprevir - India | Control - India
Number analyzed (Participants) | 47 | 23
Percentage of Participants | 53.19 | 21.74
Statistical Analysis 1: Comparison: Boceprevir - India vs Control - India; Between-Group Comparison; Test type: Superiority or Other; p = 0.0086, Miettinen and Numinen; Difference in Percentage = 33.18, 95% CI 2-sided [8.96 to 51.83]

5. Secondary Outcome: Percentage of Participants in Korea and Taiwan Achieving Early Virologic Response (EVR) at Treatment Week 8
Description: Percentage of participants achieving early virologic response (undetectable HCV-RNA at Treatment Week 8)
Time Frame: Treatment Week 8
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Boceprevir - Korea+Taiwan | Control - Korea+Taiwan
Number analyzed (Participants) | 133 | 65
Percentage of Participants | 73.68 | 44.62
Statistical Analysis 1: Comparison: Boceprevir - Korea+Taiwan vs Control - Korea+Taiwan; Between-Group Comparison; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen; Difference in Percentage = 29.08, 95% CI 2-sided [15.26 to 42.22]

6. Secondary Outcome: Percentage of Participants in India Achieving EVR at Treatment Week 8
Description: Percentage of participants achieving early virologic response (undetectable HCV-RNA at Treatment Week 8)
Time Frame: Treatment Week 8
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Boceprevir - India | Control - India
Number analyzed (Participants) | 47 | 24
Percentage of Participants | 59.57 | 25.00
Statistical Analysis 1: Comparison: Boceprevir - India vs Control - India; Between-Group Comparison; Test type: Superiority or Other; p = 0.004, Mittienen and Nurminen; Difference in Percentage = 36.13, 95% CI 2-sided [12.12 to 55.01]

7. Secondary Outcome: Percentage of Participants With an Adverse Event (AE) of Anemia in Korea and Taiwan
Description: Anemia is a condition in which the number of red blood cells or hemoglobin concentration is insufficient to meet the body's physiologic needs. This measure gives the percentage of participants who experienced an occurrence of modified World Health Organization (WHO) grade 1-4 anemia during the treatment period. A higher grade indicates a higher degree of anemia. This table summarizes the worst category observed within the period per participant per laboratory test (i.e., the lowest value for the hemotologic parameters).
Time Frame: Up to 96 weeks
Population: All Participants as Treated (APaT) - population consists of all randomized participants in Korea and Taiwan who received at least one dose of study treatment, corresponding to the study treatment they actually received. Only participants with at least one treatment value for a given laboratory test are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Boceprevir - Korea+Taiwan | Control - Korea+Taiwan
Number analyzed (Participants) | 133 | 65
Percentage of Participants
  Grade 1 (9.5 to <11 g/dL of hemoglobin) | 34.6 | 43.1
  Grade 2 (8.0 to <9.5 g/dL of hemoglobin) | 29.3 | 7.7
  Grade 3 (6.5 to <8.0 g/dL of hemoglobin) | 4.5 | 0.0
  Grade 4 (<6.5 g/dL of hemoglobin) | 0.0 | 0.0

8. Secondary Outcome: Percentage of Participants With an AE of Anemia in India
Description: Anemia is a condition in which the number of red blood cells (hemoglobin) is insufficient to meet the body's physiologic needs. This measure gives the percentage of participants who experienced an occurrence of modified WHO grade 1-4 anemia during the treatment period. A higher grade indicates a higher degree of anemia. This table summarizes the worst category observed within the period per participant per laboratory test (i.e., the lowest value for the hemotologic parameters).
Time Frame: Up to 96 weeks
Population: APaT - population consists of all randomized participants in India who received ≥ 1 dose of study treatment, corresponding to the study treatment they actually received. Only participants with at least one treatment value for a given laboratory test are included; participants who did not demonstrate GCP compliance were excluded from analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Boceprevir - India | Control - India
Number analyzed (Participants) | 47 | 24
Percentage of Participants
  Grade 1 (9.5 to <11 g/dL of hemoglobin) | 25.5 | 33.3
  Grade 2 (8.0 to <9.5 g/dL of hemoglobin) | 46.8 | 8.3
  Grade 3 (6.5 to <8.0 g/dL of hemoglobin) | 10.6 | 0
  Grade 4 (<6.5 g/dL of hemoglobin) | 0 | 0

9. Secondary Outcome: Percentage of Participants With an AE of Neutropenia in Korea and Taiwan
Description: Neutropenia is an abnormally low level of white blood cells (neutrophils). This measure gives the percentage of participants who experienced an occurrence of modified WHO grade 1-4 neutropenia during the treatment phase. A higher grade indicates a higher degree of neutropenia. This table summarizes the worst category observed within the period for each participant.
Time Frame: Up to 96 weeks
Population: APaT - population consists of all randomized participants in Korea and Taiwan who received at least one dose of study treatment, corresponding to the study treatment they actually received. Only participants with at least one treatment value for a given laboratory test are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Boceprevir - Korea+Taiwan | Control - Korea+Taiwan
Number analyzed (Participants) | 133 | 65
Percentage of Participants
  Grade 1 (1.0 to 1.5x10^9/L of neutrophils) | 30.1 | 41.5
  Grade 2 (0.75 to <1.0x10^9/L of neutrophils) | 24.8 | 20.0
  Grade 3 (0.5 to <0.75x10^9/L of neutrophils) | 22.6 | 12.3
  Grade 4 (<0.5x10^9/L of neutrophils) | 3.8 | 0.0

10. Secondary Outcome: Percentage of Participants With an AE of Neutropenia in India
Description: as for outcome 9
Time Frame: Up to 96 weeks
Population: as for outcome 8
Measure: Number; unit: Percentage of Participants
Arm/Group | Boceprevir - India | Control - India
Number analyzed (Participants) | 47 | 24
Percentage of Participants
  Grade 1 (1.0 to 1.5x10^9/L of neutrophils) | 51.1 | 29.2
  Grade 2 (0.75 to <1.0x10^9/L of neutrophils) | 12.8 | 4.2
  Grade 3 (0.5 to <0.75x10^9/L of neutrophils) | 6.4 | 0
  Grade 4 (<0.5x10^9/L of neutrophils) | 2.1 | 0

ADVERSE EVENTS:
Time Frame: Up to 96 weeks (including up to 38 weeks of follow-up)
Description: All Participants as Treated (APaT) - all randomized participants who received at least one (1) dose of study treatment. Due to lack of GCP compliance, 13 Indian participants were not included in this population.
Groups:
- Boceprevir - Korea + Taiwan; Boceprevir - India: PEG + RBV for 4 weeks followed by BOC + PEG + RBV for 32 weeks. At the Treatment Week 36 visit, participants with undetectable HCV-RNA at Treatment Weeks 8 and 12 will proceed to 36 weeks of post-treatment follow-up. Participants with detectable HCV-RNA at Treatment Week 8 and undetectable HCV-RNA at Treatment Week 12 will continue on BOC + PEG + RBV until Treatment Week 36, receive placebo + PEG + RBV until Treatment Week 48, and then proceed to 24 weeks of post-treatment follow-up. Participants with any HCV-RNA result at Treatment Week 8 and detectable HCV-RNA at Treatment Week 12 will discontinue treatment and proceed to 24 weeks of post-treatment follow-up.
- Control - Korea + Taiwan; Control - India: PEG + RBV for 4 weeks followed by BOC placebo + PEG + RBV for 44 weeks. Participants with undetectable HCV-RNA at Treatment Week 12 and at all subsequent assays will continue on placebo + PEG + RBV through Treatment Week 48 and proceed to 24 weeks of post-treatment follow-up. Participants with detectable HCV-RNA at Treatment Week 12 may roll over to Cross-Over BOC treatment beginning with Treatment Week 14.
Arm/Group | Boceprevir - Korea + Taiwan | Control - Korea + Taiwan | Boceprevir - India | Control - India
Serious Adverse Events (participants affected / at risk) | 16/133 | 3/65 | 0/47 | 2/24
Other Adverse Events (participants affected / at risk) | 131/133 | 62/65 | 44/47 | 15/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boceprevir - Korea + Taiwan (N=133) | Control - Korea + Taiwan (N=65) | Boceprevir - India (N=47) | Control - India (N=24)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infectious colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boceprevir - Korea + Taiwan (N=133) | Control - Korea + Taiwan (N=65) | Boceprevir - India (N=47) | Control - India (N=24)
Anaemia (Blood and lymphatic system disorders) | 53 (78) | 16 (23) | 14 (15) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 8 (12) | 8 (15) | 2 (3) | 1 (4)
Neutropenia (Blood and lymphatic system disorders) | 34 (58) | 17 (36) | 3 (3) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (7) | 1 (1) | 1 (1) | 1 (1)
Dry eye (Eye disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 10 (24) | 4 (4) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 10 (10) | 1 (1) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 19 (23) | 9 (10) | 1 (1) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 23 (33) | 5 (9) | 6 (6) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 9 (9) | 5 (6) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 13 (13) | 2 (2) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 9 (12) | 6 (7) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 27 (30) | 12 (13) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 11 (11) | 3 (4) | 2 (2) | 1 (1)
Asthenia (General disorders) | 14 (27) | 5 (9) | 18 (21) | 6 (6)
Chest discomfort (General disorders) | 5 (5) | 4 (4) | 0 (0) | 1 (1)
Chills (General disorders) | 4 (4) | 4 (5) | 0 (0) | 0 (0)
Fatigue (General disorders) | 36 (37) | 14 (18) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 16 (23) | 6 (18) | 2 (2) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Malaise (General disorders) | 10 (12) | 6 (10) | 2 (2) | 0 (0)
Pain (General disorders) | 6 (6) | 3 (3) | 7 (39) | 4 (18)
Pyrexia (General disorders) | 31 (54) | 14 (56) | 22 (372) | 10 (129)
Upper respiratory tract infection (Infections and infestations) | 9 (10) | 4 (4) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 4 (6) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Haemoglobin decreased (Investigations) | 23 (27) | 7 (9) | 21 (24) | 4 (6)
Neutrophil count decreased (Investigations) | 15 (25) | 8 (15) | 9 (9) | 0 (0)
Platelet count decreased (Investigations) | 16 (21) | 7 (10) | 5 (5) | 0 (0)
Reticulocyte count increased (Investigations) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Weight decreased (Investigations) | 6 (6) | 7 (8) | 6 (6) | 3 (3)
White blood cell count decreased (Investigations) | 16 (24) | 5 (6) | 3 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 34 (36) | 15 (17) | 4 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (6) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 33 (40) | 15 (17) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 43 (46) | 15 (20) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 38 (41) | 4 (4) | 9 (10) | 4 (4)
Headache (Nervous system disorders) | 40 (54) | 15 (23) | 0 (0) | 1 (4)
Hypoaesthesia (Nervous system disorders) | 7 (7) | 1 (2) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 7 (7) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 25 (28) | 11 (14) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (23) | 14 (15) | 2 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 (18) | 9 (10) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 9 (9) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 9 (12) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 33 (33) | 23 (23) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 43 (49) | 23 (27) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 22 (33) | 8 (8) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the trial without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial.